CLINICAL TRIAL: NCT05326672
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Benvitimod Cream in the Treatment of Mild to Moderate Atopic Dermatitis
Brief Title: Phase III Clinical Study of Benvitimod Cream in the Treatment of Mild to Moderate Atopic Dermatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Zhonghao Pharmaceutical (Unknown)
Responsible Party: Principal Investigator, Zhang jianzhong, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ-BWMD-2021
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Atopic Dermatitis
Keywords: Benvitimod Cream; Atopic Dermatitis; Topical Treatment
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benvitimod Cream (Experimental): Benvitimod cream, 1%, applied twice daily for 8 weeks after enrolment.
  Interventions: Drug: Benvitimod Cream
- Placebo (Placebo Comparator): Placebo, applied twice daily for 8 weeks after enrolment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benvitimod Cream — Benvitimod cream, 1%, applied twice daily for 8 weeks after enrolment.
  Arms: Benvitimod Cream
Drug: Placebo — Placebo, applied twice daily for 8 weeks after enrolment.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, multicenter, placebo-controlled clinical Phase III study to evaluate the safety and efficacy of Benvitimod cream, 1% twice daily for the treatment of mild to moderate atopic dermatitis. Approximately 240 participants with mild to moderate atopic dermatitis will be enrolled and randomly divided into two groups in a 2:1 ratio. They will use either the Benvitimod cream or placebo at the skin with atopic dermatitis for 8 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter, placebo-controlled clinical Phase III study to evaluate the safety and efficacy of Benvitimod cream, 1% twice daily for the treatment of mild to moderate atopic dermatitis. Approximately 240 participants with mild to moderate atopic dermatitis will be enrolled and randomly divided into two groups in a 2:1 ratio. They will use either the Benvitimod cream or placebo at the skin with atopic dermatitis for 8 weeks. Participants who had completed the 8-week clinical trial and were well tolerant to the drug were followed up in one-arm, long-term intermittent administration (up to 52 weeks period). In the long-term medication phase, at each visit point: ① When IGA ≥ 2, Benvitimod cream was continued to be used, twice daily. ② When IGA < 2, the drug was stopped. In the long-term follow-up, the interval of visits was 4 weeks during the medication phase and 8 weeks during the discontinuation phase.

The primary objective is to evaluate the efficacy and safety of Benvitimod cream in the treatment of mild to moderate atopic dermatitis. The primary endpoint is the proportion of participants with Investigator Global Assessment (IGA) of 0 (complete removal) or 1 (nearly complete removal) and a decrease of ≥2 points score from baseline to week 8. The study is anticipated to last from April 2022 to August 2023 with 240 participants recruited form about 20 centers in China.

All the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese Good Clinical Practice standard. The study has been approved by Institutional Review Board (IRB) and Ethics Committee (EC) in Peking University People's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of atopic dermatitis，course of disease ≥ 6 months，EASI ≤ 21 and 3% ≤ BSA ≤ 20%.
* IGA ≥ 3.
* Capable of giving written informed consent.

Exclusion Criteria:

* Skin lesions were limited to head, neck, hands and feet.
* ALT/AST ≥ 3 ULN、BUN/Cr ﹥ 1.5 ULN.
* Subjects with obvious cardiovascular, respiratory, gastrointestinal, liver, kidney, blood, neurological and psychological diseases that are unstable or not well controlled.
* Subjects have any systemic disease or other active skin disease that may affect the evaluation of the study results, or have scar, freckle, tattoo, etc. in the affected area that may affect the evaluation of skin lesions.
* Subjects with malignant neoplasms.
* Subjects with severe comorbid conditions may require systematic hormone therapy or other interventions, affect study participation or require frequent active monitoring (e.g., unstable chronic asthma).
* Subjects with definite skin infection with local bacteria, viruses and fungi.
* Subjects with mental illness or other reasons may interfere with participation in the study.
* Known to be allergic to any of the components of the drug.
* Severe hypersensitivity to food, drugs, insect venom, rubber, etc.
* Women who are pregnant, breast-feeding, or planning to become pregnant.
* Alcohol, drug abuse and known drug dependence.
* Prior to enrollment, the following treatments were used within the specified time period:

  1. External medication used within 2 weeks (e.g. glucocorticoids, calcineurin inhibitors, tacrolimus, PDE-4 inhibitors, etc.)
  2. Systemic immunotherapy used within 4 weeks (e.g., glucocorticoids, methotrexate, JAK inhibitors, cyclosporine, etc.).
  3. Received biologics for atopic dermatitis (e.g., IL-4 inhibitors, IL-13 inhibitors, etc.) within 4 weeks (or 5 half-life, whichever is longer).
  4. Received uv therapy and photochemotherapy within 4 weeks.
* Participated in clinical trials of other drugs or medical devices within 4 weeks.
* The patients who were considered unsuitable to participate in the study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Investigator Global Assessment (IGA) of 0 (complete removal) or 1 (nearly complete removal) and a decrease of ≥2 points score from Baseline to Week 8 | Week 8
  The IGA is a clinical tool for assessing the current state/severity of a participant's atopic dermatitis at a given timepoint. It is a static 6-point (0-5) morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema and induration as guidelines. Higher IGA scores represent more severe disease.

SECONDARY OUTCOMES:
Percentage decline in Eczema Area and Severity Index (EASI) score from Baseline to Week 8 | Week 8
  The EASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema, induration, excoriation, and lichenification, and the extent of %Body Surface Area (BSA) affected with atopic dermatitis.
  The 3 clinical signs are each graded on a 7-point scale (0 to 6) and the %BSA affected is scored on a 4-point scale (0 to 3) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall EASI score. Higher scores indicate more severe disease. EASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥75% improvement in Eczema Area and Severity Index (EASI) score from Baseline to Week 8 | Week 8
  The EASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema, induration, excoriation, and lichenification, and the extent of %Body Surface Area (BSA) affected with atopic dermatitis.
  The 3 clinical signs are each graded on a 7-point scale (0 to 6) and the %BSA affected is scored on a 4-point scale (0 to 3) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall EASI score. Higher scores indicate more severe disease. EASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥90% improvement in Eczema Area and Severity Index (EASI) score from Baseline to Week 8 | Week 8
  The EASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema, induration, excoriation, and lichenification, and the extent of %Body Surface Area (BSA) affected with atopic dermatitis.
  The 3 clinical signs are each graded on a 7-point scale (0 to 6) and the %BSA affected is scored on a 4-point scale (0 to 3) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall EASI score. Higher scores indicate more severe disease. EASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥50% improvement in Eczema Area and Severity Index (EASI) score from Baseline to Week 8 | Week 8
  The EASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema, induration, excoriation, and lichenification, and the extent of %Body Surface Area (BSA) affected with atopic dermatitis.
  The 3 clinical signs are each graded on a 7-point scale (0 to 6) and the %BSA affected is scored on a 4-point scale (0 to 3) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall EASI score. Higher scores indicate more severe disease. EASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥3 score improvement in Pruritus Visual Analogue Scale (VAS) from Baseline to Week 8 | Week 8
  Pruritus Visual Analogue Scale (VAS) will be used to assess severity of pruritus.
Overall EASI improvement rate and its changes with time from Baseline to Week 8 | Week 8
  The EASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema, induration, excoriation, and lichenification, and the extent of %Body Surface Area (BSA) affected with atopic dermatitis.
  The 3 clinical signs are each graded on a 7-point scale (0 to 6) and the %BSA affected is scored on a 4-point scale (0 to 3) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall EASI score. Higher scores indicate more severe disease. EASI is a static assessment made without reference to previous scores.
The average IGA decrease and its changes with time from Baseline to Week 8 | Week 8
  The IGA is a clinical tool for assessing the current state/severity of a participant's atopic dermatitis at a given timepoint. It is a static 6-point (0-5) morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema and induration as guidelines. Higher IGA scores represent more severe disease.
The average DLQI decrease and its changes with time from Baseline to Week 8 | Week 8
  The DLQI is a simple dermatology-specific 10-question validated questionnaire to assess the impact of the disease on a participant's quality of life. DLQI scores range from 0 to 30, with a higher score indicating a more impaired quality of life.
The average BSA decrease and its changes with time from Baseline to Week 8 | Week 8
  The assessment of %BSA affected is an estimate of the percentage of total involved skin with atopic dermatitis. For the purpose of clinical estimation, the total palmar surface of the participant's palm and digits may be assumed to be approximately equivalent to 1% BSA. The %BSA affected by atopic dermatitis will be evaluated (from 0% to 100%). %BSA is a static assessment made without reference to previous scores.
The average Pruritus Visual Analogue Scale (VAS) decrease and its changes with time from Baseline to Week 8 | Week 8
  Pruritus Visual Analogue Scale (VAS) will be used to assess severity of pruritus.
Proportion of participants with recurrence and the time of first recurrence of 1.0% Benvitimod cream | Week 52
  Recurrence definition: participants who have new lesions after discontinuation of Benvitimod cream, and IGA ≥2.
Proportion of participants of IGA = 0 or 1 was achieved after retreatment 8 weeks in recurrence subjects | Week 52
  Recurrence definition: participants who have new lesions after discontinuation of Benvitimod cream, and IGA ≥2.
Incidence of TEAE and SAE | Week 52
  TEAE definition: treatment emergent adverse event.
Number of recurrences in recurrence participants | Week 52
  Recurrence definition: participants who have new lesions after discontinuation of Benvitimod cream, and IGA ≥2.
Proportion of participants with ≥50% improvement in Eczema Area and Severity Index (EASI) score after retreatment 8 weeks in recurrence subjects | Week 52
  Recurrence definition: participants who have new lesions after discontinuation of Benvitimod cream, and IGA ≥2.
EASI score and IGA score decreased after retreatment 8 weeks in recurrence participants | Week 52
  The EASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema, induration, excoriation, and lichenification, and the extent of %Body Surface Area (BSA) affected with atopic dermatitis.
  The 3 clinical signs are each graded on a 7-point scale (0 to 6) and the %BSA affected is scored on a 4-point scale (0 to 3) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall EASI score. Higher scores indicate more severe disease. EASI is a static assessment made without reference to previous scores.
  The IGA is a clinical tool for assessing the current state/severity of a subject's atopic dermatitis at a given timepoint. It is a static 6-point morphological assessment of overall disease severity, as determined by the investigator, using
Incidence of AE/ADR at each visit during medication | Week 52
  AE definition: adverse event. ADR definition: adverse reaction.
Incidence of SAE and TEAE leading to discontinuation | Week 52
  SAE definition: serious adverse events. TEAE definition: treatment emergent adverse event.
Incidence of clinical abnormalities such as laboratory tests and electrocardiogram (ECG) | Week 52
  Incidence of clinical abnormalities such as laboratory tests and electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No